CLINICAL TRIAL: NCT00511199
Title: A Randomized, Open-Label, Comparative, Multi -Center Trial to Evaluate Contraceptive Efficacy, Cycle Control, Safety and Acceptability of a Monophasic Combined Oral Contraceptive (COC) Containing 2.5 mg Nomegestrol Acetate (NOMAC) and 1.5 mg Estradiol (E2), Compared to a Monophasic COC Containing 3 mg Drospirenone (DRSP) and 30 µg Ethinyl Estradiol (EE)
Brief Title: Efficacy and Safety of the Combined Oral Contraceptive (COC) NOMAC-E2 Compared to a COC Containing DRSP/EE (292001)(COMPLETED)(P05724)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P05724; Organon Protocol No. 292001
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NOMAC-E2 (Experimental): Nomegestrol Acetate (NOMAC) and Estradiol (E2), 2.5 mg NOMAC and 1.5 mg E2
  monophasic combined oral contraceptive
  Interventions: Drug: NOMAC-E2
- DRSP-EE (Active Comparator): Drospirenone (DRSP) and Ethinyl Estradiol (EE), 3 mg DRSP and 30 mcg EE monophasic combined oral contraceptive
  Interventions: Drug: DRSP-EE

INTERVENTIONS:
Drug: NOMAC-E2 — Nomegestrol Acetate and Estradiol Tablets, 2.5 mg
  NOMAC and 1.5 mg E2 taken once daily from Day 1 of menstrual period up to and including Day 28 for 13 consecutive 28-day menstrual cycles (1 year).
  Other Names: SCH 900121
  Arms: NOMAC-E2
Drug: DRSP-EE — Drospirenone and Ethinyl Estradiol Tablets, 3 mg DRSP and 30 mcg EE taken once daily from Day 1 of menstrual period up to and including Day 28 for 13 consecutive 28-day menstrual cycles (1 year).
  Other Names: SCH 900121
  Arms: DRSP-EE

SUMMARY:
The primary purpose of this study is to assess contraceptive efficacy, vaginal bleeding patterns (cycle control), general safety and acceptability of the nomegestrol acetate-estradiol (NOMAC-E2) combined oral contraceptive (COC) in a large group of women aged 18-50 years.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active women, at risk for pregnancy and not planning to use condoms.
* Women in need for contraception and willing to use an oral contraceptive (OC) for 12 months (13 cycles).
* At least 18 but not older than 50 years of age at the time of screening.
* Body mass index (BMI) of >/= 17 and </= 35.
* Good physical and mental health.
* Willing to give informed consent in writing.

Exclusion Criteria:

* Contraindications for contraceptive steroids.
* In accordance with the Summary of Product Characteristics (SmPC)/Package Insert of DRSP-EE, additional

contraindications related to the antimineralocorticoid activity of drospirenone

(conditions that predispose to hyperkalemia):

* Renal insufficiency
* Hepatic dysfunction
* Adrenal insufficiency
* An abnormal cervical smear (i.e.: dysplasia, cervical intraepithelial neoplasia [CIN],

Squamous Intraepithelial Lesion [SIL], carcinoma in situ, invasive carcinoma) at screening.

* Clinically relevant abnormal laboratory result at screening as judged by the investigator.
* Use of an injectable hormonal method of contraception; within 6 months of an injection with a 3-month duration, within 4 months of an injection with a 2-month duration, within 2 months of an injection with a 1-month duration.
* Before spontaneous menstruation has occurred following a delivery or abortion.
* Breastfeeding or within 2 months after stopping breastfeeding prior to the start of trial medication.
* Present use or use within 2 months prior to the start of the trial medication of the following drugs: phenytoin, barbiturates, primidone, carbamazepine, oxcarbazepine, topiramate, felbamate, rifampicin, nelfinavir, ritonavir, griseofulvin, ketoconazole, sex steroids (other than pre- and posttreatment contraceptive method) and herbal remedies containing Hypericum perforatum (St John's Wort).
* Administration of investigational drugs and/or participation in another clinical trial within 2 months prior to the start of the trial medication or during the trial period.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2152 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2008-04-01 (Actual); Study Completion 2008-04-01 (Actual)

REFERENCES:
- [Result] Mansour D, Verhoeven C, Sommer W, Weisberg E, Taneepanichskul S, Melis GB, Sundstrom-Poromaa I, Korver T. Efficacy and tolerability of a monophasic combined oral contraceptive containing nomegestrol acetate and 17beta-oestradiol in a 24/4 regimen, in comparison to an oral contraceptive containing ethinylestradiol and drospirenone in a 21/7 regimen. Eur J Contracept Reprod Health Care. 2011 Dec;16(6):430-43. doi: 10.3109/13625187.2011.614029. Epub 2011 Oct 13. PMID 21995590
- [Derived] Witjes H, Creinin MD, Sundstrom-Poromaa I, Martin Nguyen A, Korver T. Comparative analysis of the effects of nomegestrol acetate/17 beta-estradiol and drospirenone/ethinylestradiol on premenstrual and menstrual symptoms and dysmenorrhea. Eur J Contracept Reprod Health Care. 2015;20(4):296-307. doi: 10.3109/13625187.2015.1016154. Epub 2015 Feb 25. PMID 25712537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited participants from Europe, Asia and Australia.
Pre-assignment Details: In total, 2152 subjects were randomized, of which 1613 subjects to NOMAC-E2 and 539 subjects to DRSP-EE. A total of 2126 subjects were randomized and treated, of which 1591 subjects on NOMAC-E2 and 535 subjects on DRSP-EE.
Groups:
- NOMAC-E2: Monophasic combined oral contraceptive (COC) tablets containing 2.5 mg Nomegestrol Acetate (NOMAC) and 1.5 mg Estradiol (E2) taken once daily from Day 1 of menstrual
  period up to and including Day 28 (Days 1-24, active tablets; Days 25-28, placebo tablets) for 13 consecutive 28-day menstrual cycles (1 year).
- DRSP-EE: Monophasic COC tablets containing 3 mg Drospirenone (DRSP) and 30 mcg Ethinyl Estradiol (EE) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-21, active tablets; Days 22-28, placebo tablets) for 13 consecutive 28-day menstrual cycles (1 year).
Period: Overall Study
Arm/Group | NOMAC-E2 | DRSP-EE
Started | 1591 | 535
Completed | 1142 | 410
Not Completed | 449 | 125
Not completed — Unacceptable Vaginal Bleeding | 63 | 4
Not completed — Other Adverse Event (AE)/ Serious AE | 227 | 52
Not completed — Withdrawal of Informed Consent | 19 | 4
Not completed — Pregnancy | 6 | 3
Not completed — Pregnancy Wish | 16 | 8
Not completed — Lost to Follow-up | 40 | 17
Not completed — Other Reason | 78 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NOMAC-E2 | DRSP-EE | Total
Number analyzed (Participants) | 1591 | 535 | 2126
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (7.0) | 27.6 (7.0) | 28.0 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1591 | 535 | 2126
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of In-treatment Pregnancies (With +2 Day Window) Per 100 Woman Years of Exposure (Pearl Index)
Description: In-treatment pregnancies were pregnancies with an estimated date of conception from the day of first intake of trial medication up to and including the day of last (active or placebo) intake of trial medication extended with a maximum of two days. Each 13 cycles (28 days per cycle) of exposure constitutes a woman year. The Pearl Index was obtained by dividing the number of in-treatment pregnancies that occurred by the time (in 100 women years) that the women were under risk of becoming pregnant.
Time Frame: 1 year (13 cycles)
Population: Restricted ITT set included all participants treated except for 2 nonpregnant participants whose exposure was excluded due to limited credibility of diary data & also excluded nonpregnant participants without >= 1 cycle expected to be at risk for pregnancy (with recorded use of condoms or w/o confirmed sexual intercourse, based on e-diary data).
Measure: Number (95% Confidence Interval); unit: Pregnancies per 100 woman years
Units Other Than Participants: woman years (rounded to nearest integer)
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1442 | 486
Number analyzed (woman years (rounded to nearest integer)) | 857 | 295
Pregnancies per 100 woman years
  Overall group | 0.467 [0.1271 to 1.1948] | 1.017 [0.2097 to 2.971]
  =<35 years old (n= 1193; n=402) | 0.571 [0.1555 to 1.4614] | 1.261 [0.2601 to 3.6858]
  >35 years old (n= 249; n=84) | 0.000 [0 to 2.3594] | 0.000 [0 to 6.4466]

2. Primary Outcome: Number of In-treatment Pregnancies (With +14 Day Window) Per 100 Woman Years of Exposure (Pearl Index)
Description: In-treatment pregnancies were pregnancies with an estimated date of conception from the day of first intake of trial medication up to and including the day of last (active or placebo) intake of trial medication extended with a period of 14 days. Each 13 cycles (28 days per cycle) of exposure constitutes a woman year. The Pearl Index was obtained by dividing the number of in-treatment pregnancies that occurred by the time (in 100 women years) that the women were under risk of becoming pregnant.
Time Frame: 1 year (13 cycles)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Pregnancies per 100 woman years
Units Other Than Participants: woman years (rounded to nearest integer)
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1442 | 486
Number analyzed (woman years (rounded to nearest integer)) | 857 | 295
Pregnancies per 100 woman years
  Overall group | 0.817 [0.3283 to 1.6826] | 1.356 [0.3693 to 3.4707]
  =<35 years old (n=1193; n=402) | 0.999 [0.4016 to 2.058] | 1.682 [0.4582 to 4.3056]
  >35 years old (n=249; n=84) | 0.000 [0 to 2.3594] | 0.000 [0 to 6.4466]

3. Secondary Outcome: Number of Participants With an Occurrence of Breakthrough Bleeding/Spotting
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using e-diaries. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Breakthrough bleeding/spotting was defined as any episode that occurred during the "expected non-bleeding period" that was neither an early nor a continued withdrawal bleeding. Expected non-bleeding period: DRSP-EE group: 21-day period starting on Day 1 of the cycle; NOMAC-E2: 21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 13 cycles (one year total)
Population: The ITT group consisted of all participants who were treated; ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
  n= number of participants with evaluable cycles.
Measure: Number; unit: participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1524 | 503
participants
  Cycle 1 (n=1466 NOMAC-E2; n=470 DRSP-EE) | 483 | 130
  Cycle 2 (n=1339 NOMAC-E2; n=440 DRSP-EE) | 289 | 75
  Cycle 3 (n=1233 NOMAC-E2; n=398 DRSP-EE) | 297 | 54
  Cycle 4 (n=1135 NOMAC-E2; n=389 DRSP-EE) | 231 | 59
  Cycle 5 (n=1064 NOMAC-E2; n=368 DRSP-EE) | 221 | 62
  Cycle 6 (n=982 NOMAC-E2; n=349 DRSP-EE) | 182 | 53
  Cycle 7 (n=931 NOMAC-E2; n=320 DRSP-EE) | 165 | 45
  Cycle 8 (n=874 NOMAC-E2; n=298 DRSP-EE) | 127 | 47
  Cycle 9 (n=861 NOMAC-E2; n=295 DRSP-EE) | 129 | 47
  Cycle 10 (n=809 NOMAC-E2; n=271 DRSP-EE) | 121 | 32
  Cycle 11 (n=770 NOMAC-E2; n=277 DRSP-EE) | 125 | 29
  Cycle 12 (n=743 NOMAC-E2; n=259 DRSP-EE) | 110 | 30
  Cycle 13 (n=666 NOMAC-E2; n=241 DRSP-EE) | 94 | 33

4. Secondary Outcome: Number of Participants With an Occurrence of Absence of Withdrawal Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using e-diaries. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Absence of withdrawal bleeding was defined as no bleeding/spotting episode that began during or continued into the "expected bleeding period". Expected bleeding period: DRSP-EE group: 7-day period starting on Day 22 of the cycle; NOMAC-E2: 7-day period starting on Day 25 of the cycle and ending on Day 3 of the next cycle.
Time Frame: Every 28-day cycle for 13 cycles (one year total)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1524 | 503
participants
  Cycle 1 (n=1466 NOMAC-E2; n=470 DRSP-EE) | 284 | 14
  Cycle 2 (n=1339 NOMAC-E2; n=440 DRSP-EE) | 237 | 17
  Cycle 3 (n=1233 NOMAC-E2; n=398 DRSP-EE) | 258 | 18
  Cycle 4 (n=1135 NOMAC-E2; n=389 DRSP-EE) | 244 | 20
  Cycle 5 (n=1064 NOMAC-E2; n=368 DRSP-EE) | 245 | 17
  Cycle 6 (n=982 NOMAC-E2; n=349 DRSP-EE) | 249 | 10
  Cycle 7 (n=931 NOMAC-E2; n=320 DRSP-EE) | 245 | 11
  Cycle 8 (n=874 NOMAC-E2; n=298 DRSP-EE) | 235 | 9
  Cycle 9 (n=861 NOMAC-E2; n=295 DRSP-EE) | 245 | 13
  Cycle 10 (n=809 NOMAC-E2; n=271 DRSP-EE) | 245 | 12
  Cycle 11 (n=770 NOMAC-E2; n=277 DRSP-EE) | 232 | 17
  Cycle 12 (n=743 NOMAC-E2; n=259 DRSP-EE) | 227 | 12
  Cycle 13 (n=666 NOMAC-E2; n=241 DRSP-EE) | 279 | 14

5. Secondary Outcome: Number of Participants With an Occurrence of Breakthrough Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using e-diaries. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Breakthrough bleeding was defined as any bleeding episode that occurred during the "expected non-bleeding period" that was neither part of an early nor continued withdrawal bleeding. Expected non-bleeding period: LNG-EE group: 21-day period starting on Day 1 of the cycle; NOMAC-E2: 21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 13 cycles (one year total)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1524 | 503
Participants
  Cycle 1 (n=1466 NOMAC-E2; n=470 DRSP-EE) | 129 | 24
  Cycle 2 (n=1339 NOMAC-E2; n=440 DRSP-EE) | 63 | 20
  Cycle 3 (n=1233 NOMAC-E2; n=398 DRSP-EE) | 61 | 16
  Cycle 4 (n=1135 NOMAC-E2; n=389 DRSP-EE) | 54 | 11
  Cycle 5 (n=1064 NOMAC-E2; n=368 DRSP-EE) | 52 | 12
  Cycle 6 (n=982 NOMAC-E2; n=349 DRSP-EE) | 43 | 8
  Cycle 7 (n=931 NOMAC-E2; n=320 DRSP-EE) | 41 | 7
  Cycle 8 (n=874 NOMAC-E2; n=298 DRSP-EE) | 28 | 5
  Cycle 9 (n=861 NOMAC-E2; n=295 DRSP-EE) | 32 | 7
  Cycle 10 (n=809 NOMAC-E2; n=271 DRSP-EE) | 23 | 7
  Cycle 11 (n=770 NOMAC-E2; n=277 DRSP-EE) | 27 | 7
  Cycle 12 (n=743 NOMAC-E2; n=259 DRSP-EE) | 30 | 13
  Cycle 13 (n=666 NOMAC-E2; n=241 DRSP-EE) | 21 | 12

6. Secondary Outcome: Number of Participants With an Occurrence of Breakthrough Spotting (Spotting Only)
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using e-diaries. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Breakthrough spotting was defined as any spotting episode that occurred during the "expected non-bleeding period" that was neither part of an early nor continued withdrawal bleeding.
  Expected non-bleeding period: DRSP-EE group: 21-day period starting on Day 1 of
  the cycle; NOMAC-E2: 21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 13 cycles (one year total)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1524 | 503
Participants
  Cycle 1 (n=1466 NOMAC-E2; n=470 DRSP-EE) | 408 | 118
  Cycle 2 (n=1339 NOMAC-E2; n=440 DRSP-EE) | 244 | 58
  Cycle 3 (n=1233 NOMAC-E2; n=398 DRSP-EE) | 257 | 42
  Cycle 4 (n=1135 NOMAC-E2; n=389 DRSP-EE) | 186 | 51
  Cycle 5 (n=1064 NOMAC-E2; n=368 DRSP-EE) | 180 | 52
  Cycle 6 (n=982 NOMAC-E2; n=349 DRSP-EE) | 148 | 45
  Cycle 7 (n=931 NOMAC-E2; n=320 DRSP-EE) | 135 | 40
  Cycle 8 (n=874 NOMAC-E2; n=298 DRSP-EE) | 104 | 43
  Cycle 9 (n=861 NOMAC-E2; n=295 DRSP-EE) | 106 | 40
  Cycle 10 (n=809 NOMAC-E2; n=271 DRSP-EE) | 105 | 27
  Cycle 11 (n=770 NOMAC-E2; n=277 DRSP-EE) | 100 | 22
  Cycle 12 (n=743 NOMAC-E2; n=259 DRSP-EE) | 87 | 18
  Cycle 13 (n=666 NOMAC-E2; n=241 DRSP-EE) | 76 | 22

7. Secondary Outcome: Number of Participants With an Occurrence of Early Withdrawal Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using e-diaries. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Early withdrawal bleeding was defined as any withdrawal bleeding that started before the current "expected bleeding period". Expected bleeding period: DRSP-EE group: 7-day period starting on Day 22 of the cycle; NOMAC-E2: 7-day period starting on Day 25 of the cycle and ending on Day 3 of the next cycle.
Time Frame: Every 28-day cycle for 13 cycles (one year total)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1524 | 503
Participants
  Cycle 1 (n=1466 NOMAC-E2; n=470 DRSP-EE) | 142 | 52
  Cycle 2 (n=1339 NOMAC-E2; n=440 DRSP-EE) | 93 | 29
  Cycle 3 (n=1233 NOMAC-E2; n=398 DRSP-EE) | 80 | 22
  Cycle 4 (n=1135 NOMAC-E2; n=389 DRSP-EE) | 69 | 20
  Cycle 5 (n=1064 NOMAC-E2; n=368 DRSP-EE) | 55 | 22
  Cycle 6 (n=982 NOMAC-E2; n=349 DRSP-EE) | 34 | 16
  Cycle 7 (n=931 NOMAC-E2; n=320 DRSP-EE) | 36 | 18
  Cycle 8 (n=874 NOMAC-E2; n=298 DRSP-EE) | 31 | 12
  Cycle 9 (n=861 NOMAC-E2; n=295 DRSP-EE) | 33 | 11
  Cycle 10 (n=809 NOMAC-E2; n=271 DRSP-EE) | 19 | 9
  Cycle 11 (n=770 NOMAC-E2; n=277 DRSP-EE) | 27 | 9
  Cycle 12 (n=743 NOMAC-E2; n=259 DRSP-EE) | 18 | 9
  Cycle 13 (n=666 NOMAC-E2; n=241 DRSP-EE) | 17 | 8

8. Secondary Outcome: Number of Participants With an Occurrence of Continued Withdrawal Bleeding
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using e-diaries. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Continued withdrawal bleeding was defined as any withdrawal bleeding that continued into the "expected non-bleeding period" of the next cycle. Expected non-bleeding period: DRSP-EE group: 21-day period starting on Day 1 of the cycle; NOMAC-E2: 21-day period starting on Day 4 of the cycle.
Time Frame: Every 28-day cycle for 12 cycles
Population: The ITT group consisted of all participants who were treated; ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
Measure: Number; unit: Participants
Groups:
- NOMAC-E2: Monophasic combined oral contraceptive (COC) tablets containing 2.5 mg Nomegestrol Acetate (NOMAC) and 1.5 mg Estradiol (E2) taken once daily from Day 1 of menstrual
  period up to and including Day 28 (Days 1-24, active tablets; Days 25-28, placebo tablets) for 13 consecutive 28-day menstrual cycles (1 year).
  n= number of participants with evaluable cycles (except for the very last cycle of a participant for which this parameter was not defined).
- DRSP-EE: Monophasic COC tablets containing 3 mg Drospirenone (DRSP) and 30 mcg Ethinyl Estradiol (EE) taken once daily from Day 1 of menstrual period up to and including Day 28 (Days 1-21, active tablets; Days 22-28, placebo tablets) for 13 consecutive 28-day menstrual cycles (1 year).
  n= number of participants with evaluable cycles (except for the very last cycle of a participant for which this parameter was not defined).
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1524 | 503
Participants
  Cycle 1 (n=1455 NOMAC-E2; n=466 DRSP-EE) | 412 | 283
  Cycle 2 (n=1320 NOMAC-E2; n=437 DRSP-EE) | 406 | 274
  Cycle 3 (n=1201 NOMAC-E2; n=397 DRSP-EE) | 364 | 243
  Cycle 4 (n=1120 NOMAC-E2; n=387 DRSP-EE) | 321 | 222
  Cycle 5 (n=1051 NOMAC-E2; n=365 DRSP-EE) | 280 | 203
  Cycle 6 (n=965 NOMAC-E2; n=348 DRSP-EE) | 285 | 190
  Cycle 7 (n=920 NOMAC-E2; n=318 DRSP-EE) | 247 | 190
  Cycle 8 (n=868 NOMAC-E2; n=296 DRSP-EE) | 224 | 170
  Cycle 9 (n=854 NOMAC-E2; n=291 DRSP-EE) | 228 | 176
  Cycle 10 (n=806 NOMAC-E2; n=269 DRSP-EE) | 191 | 158
  Cycle 11 (n=766 NOMAC-E2; n=276 DRSP-EE) | 195 | 162
  Cycle 12 (n=725 NOMAC-E2; n=257 DRSP-EE) | 184 | 153

9. Secondary Outcome: Average Number of Breakthrough Bleeding/Spotting Days
Description: as for outcome 3
Time Frame: Every 28-day cycle for 13 cycles (one year total)
Population: ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
  n= number of participants who had breakthrough bleeding/spotting for the respective cycle.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1524 | 503
days
  Cycle 1 (n=483 NOMAC-E2; n=130 DRSP-EE) | 4.6 (3.6) | 4.2 (3.0)
  Cycle 2 (n=289 NOMAC-E2; n=75 DRSP-EE) | 3.5 (2.8) | 3.2 (2.5)
  Cycle 3 (n=297 NOMAC-E2; n=54 DRSP-EE) | 3.4 (2.6) | 3.6 (2.8)
  Cycle 4 (n=231 NOMAC-E2; n=59 DRSP-EE) | 3.1 (2.5) | 2.9 (2.5)
  Cycle 5 (n=221 NOMAC-E2; n=62 DRSP-EE) | 3.2 (2.5) | 2.9 (2.8)
  Cycle 6 (n=182 NOMAC-E2; n=53 DRSP-EE) | 3.3 (2.5) | 2.4 (2.0)
  Cycle 7 (n=165 NOMAC-E2; n=45 DRSP-EE) | 3.2 (2.5) | 3.0 (2.8)
  Cycle 8 (n=127 NOMAC-E2; n=47 DRSP-EE) | 3.1 (2.4) | 2.7 (1.9)
  Cycle 9 (n=129 NOMAC-E2; n=47 DRSP-EE) | 3.4 (2.6) | 2.6 (2.2)
  Cycle 10 (n=121 NOMAC-E2; n=32 DRSP-EE) | 3.1 (2.5) | 3.1 (2.6)
  Cycle 11 (n=125 NOMAC-E2; n=29 DRSP-EE) | 2.8 (2.4) | 2.6 (2.5)
  Cycle 12 (n=110 NOMAC-E2; n=30 DRSP-EE) | 3.1 (2.2) | 2.6 (2.3)
  Cycle 13 (n=94 NOMAC-E2; n=33 DRSP-EE) | 2.7 (2.0) | 3.2 (2.6)

10. Secondary Outcome: Average Number of Withdrawal Bleeding/Spotting Days
Description: Cycle control was evaluated on the basis of vaginal bleeding pattern as recorded daily by participants using e-diaries. Participants documented whether vaginal bleeding was present, and if present, indicated whether it was considered to be spotting or bleeding. Withdrawal bleeding was defined as bleeding/spotting episode that started during or continued into the "expected bleeding period". Expected bleeding period: DRSP-EE group: 7-day period starting on Day 22 of the cycle; NOMAC-E2: 7-day period starting on Day 25 of the cycle and ending on Day 3 of the next cycle.
Time Frame: Every 28-day cycle for 13 cycles (one year total)
Population: ITT analyses of vaginal bleeding patterns were based on all participants in the ITT group who had at least one evaluable cycle. Cycles were considered to be non-evaluable in case of insufficient bleeding data or improper cycle length.
  n= number of participants who had withdrawal bleeding/spotting for the respective cycle.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NOMAC-E2 | DRSP-EE
Number analyzed (Participants) | 1524 | 503
days
  Cycle 1 (n=1182 NOMAC-E2; n=456 DRSP-EE) | 5.7 (11.2) | 6.0 (3.3)
  Cycle 2 (n=1102 NOMAC-E2; n=423 DRSP-EE) | 5.6 (15.1) | 5.5 (2.2)
  Cycle 3 (n=975 NOMAC-E2; n=380 DRSP-EE) | 5.9 (19.0) | 5.4 (2.4)
  Cycle 4 (n=891 NOMAC-E2; n=369 DRSP-EE) | 6.0 (19.9) | 5.4 (3.5)
  Cycle 5 (n=819 NOMAC-E2; n=351 DRSP-EE) | 6.0 (20.8) | 5.3 (3.4)
  Cycle 6 (n=733 NOMAC-E2; n=339 DRSP-EE) | 5.8 (21.8) | 5.2 (2.8)
  Cycle 7 (n=686 NOMAC-E2; n=309 DRSP-EE) | 5.8 (22.4) | 5.2 (2.5)
  Cycle 8 (n=639 NOMAC-E2; n=289 DRSP-EE) | 5.6 (22.3) | 5.7 (8.5)
  Cycle 9 (n=616 NOMAC-E2; n=282 DRSP-EE) | 5.7 (21.9) | 5.7 (8.5)
  Cycle 10 (n=564 NOMAC-E2; n=259 DRSP-EE) | 5.7 (23.5) | 5.5 (8.2)
  Cycle 11 (n=538 NOMAC-E2; n=260 DRSP-EE) | 6.0 (24.1) | 5.6 (8.3)
  Cycle 12 (n=516 NOMAC-E2; n=247 DRSP-EE) | 5.6 (21.3) | 5.7 (8.9)
  Cycle 13 (n=387 NOMAC-E2; n=227 DRSP-EE) | 4.9 (23.9) | 4.2 (3.8)

ADVERSE EVENTS:
Arm/Group | NOMAC-E2 | DRSP-EE
Serious Adverse Events (participants affected / at risk) | 38/1591 | 13/535
Other Adverse Events (participants affected / at risk) | 849/1591 | 242/535
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOMAC-E2 (N=1591) | DRSP-EE (N=535)
Vestibular neuronitis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cryptosporidiosis infection (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis viral (Infections and infestations) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0)
Giardiasis (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 2 (2) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Multiple Sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Haematosalpinx (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOMAC-E2 (N=1591) | DRSP-EE (N=535)
Influenza (Infections and infestations) | 55 (61) | 30 (36)
Nasopharyngitis (Infections and infestations) | 144 (190) | 53 (66)
Vaginal candidiasis (Infections and infestations) | 127 (143) | 45 (53)
Weight increased (Investigations) | 158 (162) | 37 (38)
Headache (Nervous system disorders) | 217 (405) | 72 (123)
Cervical dysplasia (Reproductive system and breast disorders) | 111 (112) | 39 (40)
Withdrawal bleeding irregular (Reproductive system and breast disorders) | 188 (424) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 280 (335) | 47 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR recognizes the right of the investigator(s) to publish, but all publications must be based on data validated and released by the SPONSOR. Any such scientific paper, presentation, or other communication concerning the clinical trial will first be submitted to the SPONSOR, at least six weeks ahead of estimated publication or presentation, for consent, which shall not be withheld unreasonably.